CLINICAL TRIAL: NCT06526039
Title: A Short Regimen for Patients With Rifampicin-resistant Isoniazid-susceptible Tuberculosis
Brief Title: A Short Regimen for Rifampicin-resistant Isoniazid-susceptible TB
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Hualien Tzu Chi General Hospital (Other); Chest Hospital, Ministry of Health and Welfare, Taiwan (Other Government); Chang-Hua Hospital (Other Government); Taichung Veterans General Hospital (Other); Taichung Hospital, Ministry of Health and Welfare (Unknown); Taoyuan General Hospital (Other Government); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chen-Yuan Chiang, Vice superintendent, Taipei Medical University WanFang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N202404036
Record Dates: First submitted 2024-07-10; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Tuberculosis, Pulmonary
Keywords: bedaquiline; isoniazid; moxifloxacin; tuberculosis; rifampicin resistance
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Patients will be treated with a novel short regimen
  Interventions: Other: a novel short regimen

INTERVENTIONS:
Other: a novel short regimen — An intensive phase consisting of isoniazid, bedaquiline, moxifloxacin and pyrazinamide for 2 months (9 weeks). A continuation phase consisting of isoniazid, bedaquiline, and levofloxacin for 4 months (17 weeks). Treatment may be extended for 3 months (13 weeks) in patients with severe disease or with delayed culture conversion, defined by culture positive at 4 months of treatment.

SUMMARY:
To assess outcome of treatment and safety among patients with rifampicin-resistant isoniazid-susceptible pulmonary tuberculosis treated with a novel regimen consisting of isoniazid, bedaquiline, and moxifloxacin throughout for 6 months, supplemented by pyrazinamide for the initial 2 months.

DETAILED DESCRIPTION:
Rifampicin-resistant tuberculosis (RR-TB) could be classified into rifampicin-resistant, isoniazid-susceptible TB (RrHs-TB) and rifampicin-resistant, isoniazid-resistant TB (MDR-TB), that is MDR-TB. RrHs-TB and MDR-TB are different because isoniazid has potent early bactericidal activity (EBA) and remains susceptible in RrHs-TB.

The standard first line anti-TB regimen recommended by WHO consisting of isoniazid and rifampicin throughout for 6 months supplemented by pyrazinamide and ethambutol for the initial 2 months (2HRZE/4HR). The duration of treatment of the first line standard 6-month regimen is mainly determined by the sterilization power of the core drug, namely rifampicin, paired with pyrazinamide. Moxifloxacin had potent EBA that is comparable to that of isoniazid. Bedaquiline has delayed onset of action but after a few days of treatment its EBA is comparable to that of isoniazid and rifampicin. Both moxifloxacin and bedaquiline have potent sterilizing activity.

To avoid the use of a toxic MDR-TB regimen, we hypothesize that the combination of bedaquiline and moxifloxacin is non inferior to rifampicin in terms of EBA and sterilizing activity, and could be used to substitute for rifampicin in the standard first line anti-TB regimen (2HRZE/4HR) as a novel approach for the treatment of RrHs-TB, as well as TB patients for whom rifamycin is intolerable (Ri-TB) and TB patients for whom rifamycin-sparing anti-TB regimens are preferred due to drug-drug interaction (Rs-TB).

Trial intervention

The novel regimen will be given in two phases:

1. An intensive phase consisting of isoniazid, bedaquiline, moxifloxacin and pyrazinamide for 2 months (9 weeks). Exclusion of isoniazid resistance by conventional phenotypic method or by a rapid molecular test before treatment initiation is required. Amikacin will be added before obtaining results of conventional DST if exclusion of isoniazid resistance is done by a molecular test at treatment initiation. If isoniazid resistance is again excluded by a repeat molecular test (either the same or a different molecular test), amikacin could be dropped after two weeks of treatment.
2. A continuation phase consisting of isoniazid, bedaquiline, and levofloxacin for 4 months (17 weeks). Treatment may be extended for 3 months (13 weeks) in patients with severe disease or with delayed culture conversion, defined by culture positive at 4 months of treatment. If pyrazinamide is discontinued earlier due to adverse reaction, the continuation phase will be extended for 3 months (13 weeks) for a total treatment duration of 9 months (39 weeks).

Selection of patients

The target population is:

1. Patients diagnosed with rifampicin-resistant isoniazid-susceptible TB (RrHs-TB),

   The following two type of patients will also be enrolled because rifamycin will not be used in the treatment of TB
2. Patients diagnosed with susceptible TB who are not able to tolerate rifampicin due to adverse reactions, in whom rifabutin is intolerable or clinically not indicated (Ri-TB),
3. Patients with TB for whom rifampicin-sparing anti-TB regimens is preferred (such as organ transplant recipients) due to drug-drug interaction (Rs-TB).

Type of design

This is a prospective open-label single-group study that participants will be treated with a novel regimen.

Trial objectives

The primary objectives of the trial are:

1. To assess the proportion of patients with a favourable efficacy outcome on the study regimen.
2. To assess the proportion of patients who experience grade 3 or greater adverse events during treatment and follow-up in the study regimen.

Outcome measures

The primary efficacy outcome measure is the proportion of patients with a favourable outcome at 12 months (53 weeks) post treatment initiation.

A patient's outcome will be classified as favourable if they have a negative culture result 12 months (53 weeks) after treatment initiation not having been previously classified as unfavourable.

A patient's outcome will be classified as unfavourable if:

1. they are discontinued from their allocated study treatment and subsequently restarted on a different regimen,
2. treatment is extended beyond the scheduled end of treatment for any reason other than making up of missed treatment,
3. they are restarted on any MDR-TB treatment after the scheduled end of treatment,
4. they change their allocated study treatment for any reason other than the replacement of a single drug,
5. they die at any point up to 12 months post treatment initiation,
6. they have a positive culture result at 12 months post treatment initiation.

The primary safety outcome measure is the proportion of patients experiencing a grade 3 or greater adverse event, as defined by the CTCAE criteria except hyperuricemia which will be defined by the DAIDS criteria, during treatment and follow-up to 12 months (53 weeks) post treatment initiation.

Secondary outcome measures include:

* Time to sputum (smear and culture) conversion
* Time to unfavourable efficacy outcome
* The proportion of patients with a favourable outcomes at 24 months post treatment initiation
* All causes mortality during treatment and follow-up
* The proportion of patients with a change of 2 or more drugs for adverse drug reactions
* Number of adverse reactions occurring on treatment
* The proportion of patients with treatment interruption for 2 or months

Sample Size

We adopt the approach of the Nix-TB study and the ZeNix trial and hypothesize that the proportion of patients with favourable efficacy outcomes at 12 months (53 weeks) after treatment initiation would be greater than 50%. The trial does not have a control group. A sample of 45 participants would provide more than 90% power to demonstrate that the lower boundary of the 95% confidence interval is greater than 50%, using a two-sided 5% significance level. We plan to expand the enrollment to at least 80 patients to assess the primary efficacy of the study regimen.

Analysis population definitions

Intention-to-treat (ITT)

All enrolled patients will be included in the ITT analysis population.

Safety population

All patients who have taken at least one dose of trial treatment will be included in the safety analysis population.

Modified intention-to-treat (mITT)

The mITT population is defined as all enrolled patients that have a positive culture for M. tuberculosis on LJ or MGIT media at screening, with the exception of rifampicin-resistant isoniazid susceptible TB patients with isolates taken before treatment initiation that are subsequently found to be susceptible to rifampicin, and patients with isolates taken before treatment initiation that are subsequently found to be resistant to fluoroquinolones on phenotypic DST. Whole genome sequencing will be done for strains with discordant results between phenotypic and genotypic methods. Results from the national reference mycobacteriology laboratory of Taiwan CDC will take priority over any results from local laboratories where available.

Per protocol (PP)

The PP population will be the same as the mITT population with the exclusion of patients not completing a protocol-adherent course of treatment, other than for treatment failure or death. Treatment failure is defined as failure to attain and maintain culture negativity until the end of allocated treatment.

Definition of a protocol-adherent course of treatment

Patients will be excluded from the per-protocol analysis if they do not complete a protocol adherent course of treatment, other than for treatment failure or death.

A patient will have completed a protocol-adherent course of treatment when they have taken 80% of doses within 120% of the minimum duration in both the intensive phase and in the whole treatment period. For this purpose, a dose is defined as all the study medications at the correct dose for that particular day.

For the study Regimen, with or without an extension, a patient will have completed a protocol-adherent course of treatment if they have taken:

* 50 doses (80% of 9 weeks) within 76 days (120% of 9 weeks) in the intensive phase, and
* 157 doses (80% of 28 weeks) within 235 days (120% of 28 weeks) over the whole treatment period (i.e. the combined intensive and continuation phases) regardless of treatment extensions.

Statistical significance

P value <0.05 will be considered statistically significant in this trial.

ELIGIBILITY:
Inclusion Criteria:

A patient will be eligible for entry to the study if he/she:

* Is willing and able to give informed consent to be enrolled in the trial treatment and follow-up (signed or witnessed consent if the patient is illiterate)
* Is aged 18 years or older
* Has bacteriologically-confirmed pulmonary tuberculosis by Xpert MTB/RIF, other nucleic acid amplification test, or culture
* With initial laboratory result of resistance to rifampicin by Xpert MTB/RIF or Xpert MTB/RIF ultra, or other DST (line probe assay, culture); and with initial laboratory result that is susceptible to isoniazid by Xpert MTB/RIF or other DST. If rifampicin resistance is detected by Xpert MTB/RIF or Xpert MTB/RIF ultra in specimens with very low bacillary, rifampicin resistance has been confirmed by a repeat molecular test.
* With initial laboratory result of being susceptible to rifampicin by Xpert MTB/RIF or other DST (Xpert MTB/RIF ultra, line probe assay, culture) but are not able to tolerate rifampicin for whom rifabutin is intolerable or clinically not indicated; and with initial laboratory result that is susceptible to isoniazid by Xpert MTB/RIF or other DST
* With initial laboratory result of being susceptible to rifampicin by Xpert MTB/RIF or other DST (Xpert MTB/RIF ultra, line probe assay, culture) but rifamycin-sparing regimens are preferred due to drug-drug interaction, such as organ transplant recipients; and with initial laboratory result that is susceptible to isoniazid by Xpert MTB/RIF or other DST.
* With initial laboratory result that is susceptible to fluoroquinolone by Xpert MTB/XDR or other DST.
* If HIV test positive, is willing to be treated with ART in accordance with the national policies.
* Agrees to use effective barrier contraception or have an intrauterine contraceptive device during treatment phase if a pre-menopausal woman
* Has an identifiable address and expects to remain in the area for the duration of the study
* Is willing to adhere to the follow-up schedule and to study procedures

Exclusion Criteria:

A patient will not be eligible for entry to the study if he/she:

* Is infected with a strain of M. Tuberculosis resistant to isoniazid by Xpert MTB/XDR or other tests
* Is infected with a strain of M. Tuberculosis resistant to fluoroquinolone by Xpert MTB/XDR or other tests
* Is infected with a strain of M. Tuberculosis resistant to amikacin by Xpert MTB/XDR or other tests and have no result of susceptibility of isoniazid by conventional drug susceptibility testing
* Has tuberculous meningitis or bone and joint tuberculosis
* Is critically ill, and in the judgment of the investigator, unlikely to survive more than 4 months.
* Is known to be pregnant or breast-feeding
* Is unable to attend or comply with treatment or follow-up schedule
* Is unable to take oral medication
* Has AST or ALT >5 times the upper limit of normal
* Has AST or ALT > 3 times the upper limit of normal ,and either with symptoms of hepatitis or bilirubin > 1.5 times the upper limit of normal
* Has any condition (social or medical) which in the opinion of the investigator would make study participation unsafe.
* Is taking any medications contraindicated with the medicines in either the trial or control regimen
* Has a known allergy to any fluoroquinolone antibiotic
* Is currently taking part in another trial of a medicinal product
* Has a QTcF interval of ≥450msec at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with a favourable outcome at 12 months (53 weeks) post treatment initiation | 12 months after treatment initiation
  The primary efficacy outcome measure is the proportion of patients with a favourable outcome at 12 months (53 weeks) post treatment initiation
the proportion of patients experiencing a grade 3 or greater adverse event during treatment and follow-up to 12 months (53 weeks) post treatment initiation. | from treatment initiation to 12 months after treatment initiation
  The primary safety outcome measure is the proportion of patients experiencing a grade 3 or greater adverse event, as defined by the CTCAE criteria except hyperuricemia which will be defined by the DAIDS criteria, during treatment and follow-up to 12 months (53 weeks) post treatment initiation.

SECONDARY OUTCOMES:
Sputum conversion | through study completion, an average of 9 months
  Time to sputum (smear and culture) conversion
Time to unfavourable efficacy outcome | through study completion, an average of 9 months
  A patient's outcome will be classified as unfavourable if:
  1. they are discontinued from their allocated study treatment and subsequently restarted on a different regimen,
  2. treatment is extended beyond the scheduled end of treatment for any reason other than making up of missed treatment,
  3. they are restarted on any MDR-TB treatment after the scheduled end of treatment,
  4. they change their allocated study treatment for any reason other than the replacement of a single drug,
  5. they die at any point up to 12 months post treatment initiation,
  6. they have a positive culture result at 12 months post treatment initiation.
the proportion of patients with a favourable outcome at 24 months (105 weeks) post treatment initiation | from treatment initiation to 24 months after treatment initiation
  The secondary efficacy outcome measure is the proportion of patients with a favourable outcome at 24 months (105 weeks) post treatment initiation.
mortality during treatment and follow-up | from treatment initiation to 24 months after treatment initiation
  All cause mortality during treatment and follow-up
Change of regimen for adverse drug reactions | through study completion, an average of 9 months
  The proportion of patients with a change of two or more drugs for adverse drug reactions
Number of adverse drug reactions | through study completion, an average of 9 months
  The number of adverse drug reactions occurring on treatment
Proportion of patients with treatment interruption for 2 months | through study completion, an average of 9 months
  The proportion of patients with treatment interruption for 2 or more months